CLINICAL TRIAL: NCT00500682
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study of AST-120 for Prevention of Chronic Kidney Disease Progression in Patients With Moderate to Severe Chronic Kidney Disease
Brief Title: A Study of AST-120 for Evaluating Prevention of Progression In Chronic Kidney Disease (EPPIC-1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Kureha Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KRM-306
Record Dates: First submitted 2007-07-11; First posted 2007-07-13 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AST-120 (Experimental)
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: Placebo — 9g /day (3 times a day)
  Arms: Placebo
Drug: AST-120 — 9g /day (3 times a day)
  Arms: AST-120

SUMMARY:
1) To evaluate the effectiveness of AST-120 (spherical carbon adsorbent) added to standard-of-care therapy in moderate to severe Chronic Kidney Disease (CKD), on time to first occurrence of any event of the triple composite outcome of initiation of dialysis, kidney transplant or doubling of serum creatinine (sCr) when compared with placebo; 2) To evaluate the safety and tolerability of long-term AST-120 therapy in patients with CKD; 3) To evaluate the effects of AST-120 versus placebo, on other measures of renal function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Moderate to severe CKD, not anticipated to require dialysis or renal transplant within the next 6 months
* Patient survival expected to be no less than one year
* Serum creatinine in men >= 2.0 mg/dL (>= 177 µmol/L) and <= 5.0 mg/dL (<= 442 µmol/L), and in women >= 1.5 mg/dL (>= 133 µmol/L) and <= 5.0 mg/dL (<= 442 µmol/L) at Screening
* Urinary total protein to urinary total creatinine ratio must be >= 0.5 on a spot void at Screening
* Blood pressure <= 160/90 mmHg at both Screening and Baseline. In addition, blood pressure, if measured, must have been stable in hypertensive patients over the 3 months prior to Screening, with no more than 1 blood pressure reading > 160/90 mmHg
* In patients being treated for hypertension, they should be on a stable anti-hypertensive regimen

Exclusion Criteria:

* Obstructive or reversible cause of kidney disease
* Nephrotic syndrome defined as a ratio of urinary total protein to urinary creatinine of > 6.0 as measured on a spot void
* Adult polycystic kidney disease
* History of previous kidney transplant
* History of recent (within the past 6 months) accelerated or malignant hypertension
* Uncontrolled arrhythmia or severe cardiac disease within the past 6 months
* History of malabsorption, inflammatory bowel disease, hiatal hernia, active peptic ulcer, or severe GI dysmotility, not attributable to the use of a phosphate binder
* Received any investigational agent or participated in a clinical study within the previous 3 months
* Presence of any significant medical condition that might create an undue risk with study participation, or significantly confound the collection of safety and efficacy data in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2007-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Tanabe Pharma Development America, Inc.
Locations (105):
- United States (41):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Alhambra, California
  - Covina, California
  - Glendale, California
  - Los Angeles, California
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Hudson, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Spring Hill, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Ypsilanti, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Camden, New Jersey
  - Eatontown, New Jersey
  - Port Washington, New York
  - Springfield Gardens, New York
  - Asheville, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Rock Hill, South Carolina
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Appleton, Wisconsin
  - Oshkosh, Wisconsin
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - San Luis
  - San Miguel de Tucumán
  - San Pedro
- Brazil (7):
  - Barao Geraldo-Campinas
  - Belo Horizonte Minas Gerais
  - Juiz de Fora
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
  - Taubaté
- Canada (7):
  - Winnipeg, Manitoba
  - Brampton, Ontario
  - Kitzhener, Ontario
  - Oakville, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (5):
  - České Budějovice
  - Jihlava
  - Ostrava - Poruba
  - Prague
  - Tábor
- France (4):
  - Grenoble
  - Lyon
  - Nantes
  - Saint-Lô
- Italy (4):
  - Bologna
  - Brescia
  - Como
  - Pavia
- Mexico (3):
  - Aguascalientes
  - Mexico City
  - Tijuana
- Poland (4):
  - Gdansk
  - Szczecin
  - Torun
  - Warsaw
- Caguas, Puerto Rico
- Russia (14):
  - Bamaul
  - Kazan'
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Pyatigorsk
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Sochi
  - Stavropol
  - Yekaterinburg
- Ukraine (10):
  - Chernivtsi
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Odesa
  - Uzhhorod
  - Vinnitsa
  - Zhytomyr

REFERENCES:
- [Result] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Arita K, Kato A, Shimizu M. Randomized Placebo-Controlled EPPIC Trials of AST-120 in CKD. J Am Soc Nephrol. 2015 Jul;26(7):1732-46. doi: 10.1681/ASN.2014010042. Epub 2014 Oct 27. PMID 25349205
- [Derived] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Shimizu M, Kikuchi M, Shobu Y. Risk factors for progression of chronic kidney disease in the EPPIC trials and the effect of AST-120. Clin Exp Nephrol. 2018 Apr;22(2):299-308. doi: 10.1007/s10157-017-1447-0. Epub 2017 Jul 24. PMID 28741050
- [Derived] Schulman G, Berl T, Beck GJ, Remuzzi G, Ritz E, Shimizu M, Shobu Y, Kikuchi M. The effects of AST-120 on chronic kidney disease progression in the United States of America: a post hoc subgroup analysis of randomized controlled trials. BMC Nephrol. 2016 Sep 30;17(1):141. doi: 10.1186/s12882-016-0357-9. PMID 27716149

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AST-120 | Placebo
Started | 510 | 510
Completed | 204 | 223
Not Completed | 306 | 287
Not completed — Adverse Event | 37 | 29
Not completed — Death | 25 | 16
Not completed — Lost to Follow-up | 11 | 11
Not completed — Physician Decision | 6 | 10
Not completed — Pregnancy | 2 | 0
Not completed — Protocol Violation | 1 | 3
Not completed — Withdrawal by Subject | 80 | 74
Not completed — Reaching endpoints, Noncompliance, etc | 144 | 144

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AST-120 | Placebo | Total
Number analyzed (Participants) | 510 | 510 | 1020
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.93) | 55.8 (14.99) | 56.1 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 179 | 374
  Male | 315 | 331 | 646

OUTCOME MEASURES:

1. Primary Outcome: Composite of Dialysis Initiation, Kidney Transplantation, and Serum Creatinine Doubling. Number of Participants Meeting the Criteria Are Reported.
Time Frame: Beyond Week 48, a 12-week visit cycle continued until the end of the study or until individual patients reached an endpoint
Population: ITT (censored at last contact)
Measure: Number; unit: participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 500 | 502
participants | 178 | 177

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events and Treatment-emergent Serious Adverse Events
Time Frame: Approximately 42 months
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
Participants
  Treatment-emergent AE | 436 | 448
  Treatment-emergent SAE | 195 | 184

3. Secondary Outcome: Number of Participants Who Developed a Component of a Quadruple Composite Endpoint (Initiation of Dialysis, Kidney Transplant, Doubling of sCr, or Death)
Time Frame: Approximately 42 months
Population: ITT (censored at last contact)
Measure: Count of Participants; unit: Participants
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 500 | 502
Participants | 213 | 201

4. Secondary Outcome: Vitamin A Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, Early Term/Discontinuation (Mean: 428.615 Days), Final Visit (Mean: 947.354 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
ng/mL
  Baseline: number analyzed (Participants) | 459 | 465
  Baseline | 1145.3 (356.67) | 1164.2 (387.08)
  Week 12: number analyzed (Participants) | 432 | 438
  Week 12 | 1142.4 (374.14) | 1177.9 (404.21)
  Week 24: number analyzed (Participants) | 416 | 415
  Week 24 | 1151.5 (382.40) | 1193.6 (363.36)
  Week 36: number analyzed (Participants) | 394 | 387
  Week 36 | 1148.1 (385.90) | 1215.1 (406.78)
  Week 48: number analyzed (Participants) | 365 | 361
  Week 48 | 1156.2 (367.71) | 1210.1 (396.91)
  Week 60: number analyzed (Participants) | 342 | 346
  Week 60 | 1199.2 (388.36) | 1232.1 (419.86)
  Week 72: number analyzed (Participants) | 312 | 314
  Week 72 | 1216.0 (368.58) | 1265.5 (428.28)
  Week 84: number analyzed (Participants) | 286 | 295
  Week 84 | 1252.1 (406.11) | 1292.8 (435.80)
  Week 96: number analyzed (Participants) | 258 | 269
  Week 96 | 1240.2 (367.21) | 1314.8 (433.70)
  Week 108: number analyzed (Participants) | 202 | 212
  Week 108 | 1222.1 (367.46) | 1305.7 (421.64)
  Week 120: number analyzed (Participants) | 149 | 157
  Week 120 | 1188.8 (357.58) | 1234.7 (397.81)
  Week 132: number analyzed (Participants) | 99 | 111
  Week 132 | 1273.5 (416.43) | 1284.1 (411.37)
  Week 144: number analyzed (Participants) | 64 | 73
  Week 144 | 1305.0 (379.81) | 1277.9 (336.23)
  Week 156: number analyzed (Participants) | 41 | 52
  Week 156 | 1255.6 (323.72) | 1174.8 (347.46)
  Week 168: number analyzed (Participants) | 21 | 28
  Week 168 | 1244.6 (275.57) | 1185.9 (402.00)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 1176.5 (342.14) | 1203.5 (271.98)
  Week 192: number analyzed (Participants) | 3 | 4
  Week 192 | 1253.0 (340.63) | 1189.3 (152.33)
  Early Term/Discontinuation: number analyzed (Participants) | 135 | 130
  Early Term/Discontinuation | 1167.2 (401.08) | 1191.4 (457.79)
  Final Visit: number analyzed (Participants) | 198 | 215
  Final Visit | 1266.9 (357.06) | 1320.1 (444.09)

5. Secondary Outcome: Vitamin B12 Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, Early Term/Discontinuation (Mean: 428.114 Days), Final Visit (Mean: 947.239 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
pg/mL
  Baseline: number analyzed (Participants) | 498 | 493
  Baseline | 688.1 (1881.58) | 620.5 (1630.87)
  Week 12: number analyzed (Participants) | 449 | 458
  Week 12 | 597.3 (1824.74) | 570.0 (1347.75)
  Week 24: number analyzed (Participants) | 421 | 420
  Week 24 | 554.2 (1654.52) | 483.7 (536.30)
  Week 36: number analyzed (Participants) | 384 | 389
  Week 36 | 500.6 (568.44) | 581.6 (1316.46)
  Week 48: number analyzed (Participants) | 359 | 353
  Week 48 | 530.6 (759.54) | 500.2 (940.36)
  Week 60: number analyzed (Participants) | 331 | 339
  Week 60 | 494.2 (534.92) | 704.9 (2338.15)
  Week 72: number analyzed (Participants) | 300 | 312
  Week 72 | 545.9 (1268.50) | 661.8 (2014.14)
  Week 84: number analyzed (Participants) | 281 | 294
  Week 84 | 497.6 (923.15) | 543.1 (1246.14)
  Week 96: number analyzed (Participants) | 254 | 260
  Week 96 | 646.6 (2012.14) | 799.6 (2767.12)
  Week 108: number analyzed (Participants) | 203 | 211
  Week 108 | 544.1 (1564.38) | 682.2 (1947.45)
  Week 120: number analyzed (Participants) | 146 | 156
  Week 120 | 590.0 (1968.53) | 638.4 (1993.90)
  Week 132: number analyzed (Participants) | 98 | 111
  Week 132 | 923.7 (3358.51) | 714.2 (2262.71)
  Week 144: number analyzed (Participants) | 62 | 73
  Week 144 | 460.5 (291.19) | 472.6 (283.43)
  Week 156: number analyzed (Participants) | 41 | 51
  Week 156 | 476.3 (285.02) | 586.3 (811.97)
  Week 168: number analyzed (Participants) | 21 | 28
  Week 168 | 563.9 (528.25) | 493.7 (342.53)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 564.2 (254.57) | 653.8 (694.69)
  Week 192: number analyzed (Participants) | 3 | 4
  Week 192 | 489.0 (306.00) | 974.0 (898.28)
  Early Term/Discontinuation: number analyzed (Participants) | 134 | 130
  Early Term/Discontinuation | 935.7 (2400.94) | 953.5 (2914.40)
  Final Visit: number analyzed (Participants) | 199 | 216
  Final Visit | 626.7 (1464.99) | 747.1 (2495.49)

6. Secondary Outcome: 25-Hydroxyvitamin D Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, Early Term/Discontinuation (Mean: 427.270 Days), Final Visit (Mean: 946.762 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
ng/mL
  Baseline: number analyzed (Participants) | 505 | 503
  Baseline | 22.08 (10.361) | 22.06 (10.400)
  Week 12: number analyzed (Participants) | 463 | 462
  Week 12 | 21.55 (9.988) | 22.15 (10.162)
  Week 24: number analyzed (Participants) | 432 | 426
  Week 24 | 21.41 (9.823) | 22.13 (9.648)
  Week 36: number analyzed (Participants) | 393 | 393
  Week 36 | 21.70 (10.539) | 21.70 (9.926)
  Week 48: number analyzed (Participants) | 369 | 363
  Week 48 | 21.83 (10.963) | 22.06 (10.644)
  Week 60: number analyzed (Participants) | 343 | 346
  Week 60 | 21.78 (11.076) | 21.56 (10.425)
  Week 72: number analyzed (Participants) | 315 | 316
  Week 72 | 22.23 (10.988) | 22.29 (9.617)
  Week 84: number analyzed (Participants) | 284 | 298
  Week 84 | 21.79 (10.759) | 22.75 (10.528)
  Week 96: number analyzed (Participants) | 260 | 267
  Week 96 | 22.18 (11.563) | 22.53 (10.833)
  Week 108: number analyzed (Participants) | 203 | 213
  Week 108 | 21.85 (11.324) | 21.62 (10.679)
  Week 120: number analyzed (Participants) | 149 | 159
  Week 120 | 22.15 (11.189) | 22.45 (9.344)
  Week 132: number analyzed (Participants) | 100 | 111
  Week 132 | 22.04 (10.581) | 21.83 (10.285)
  Week 144: number analyzed (Participants) | 64 | 74
  Week 144 | 23.29 (11.051) | 22.95 (11.046)
  Week 156: number analyzed (Participants) | 41 | 52
  Week 156 | 23.23 (9.857) | 23.01 (12.943)
  Week 168: number analyzed (Participants) | 21 | 27
  Week 168 | 25.45 (12.045) | 24.44 (11.403)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 29.58 (12.985) | 28.10 (10.929)
  Week 192: number analyzed (Participants) | 3 | 4
  Week 192 | 33.10 (6.651) | 31.38 (9.606)
  Early Term/Discontinuation: number analyzed (Participants) | 137 | 133
  Early Term/Discontinuation | 20.57 (9.958) | 22.52 (11.803)
  Final Visit: number analyzed (Participants) | 199 | 217
  Final Visit | 25.20 (10.847) | 25.69 (9.937)

7. Secondary Outcome: Vitamin E Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, 192, Early Term/Discontinuation (Mean: 428.056 Days), Final Visit (Mean: 946.525 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
ug/mL
  Baseline: number analyzed (Participants) | 496 | 491
  Baseline | 17.49 (7.554) | 16.95 (6.923)
  Week 12: number analyzed (Participants) | 458 | 456
  Week 12 | 17.30 (6.880) | 16.44 (6.080)
  Week 24: number analyzed (Participants) | 422 | 419
  Week 24 | 17.55 (7.237) | 17.08 (6.560)
  Week 36: number analyzed (Participants) | 394 | 390
  Week 36 | 17.42 (6.474) | 17.22 (6.445)
  Week 48: number analyzed (Participants) | 367 | 362
  Week 48 | 17.58 (7.040) | 17.31 (6.544)
  Week 60: number analyzed (Participants) | 341 | 348
  Week 60 | 17.77 (7.376) | 17.70 (6.880)
  Week 72: number analyzed (Participants) | 313 | 315
  Week 72 | 17.50 (6.683) | 17.07 (6.119)
  Week 84: number analyzed (Participants) | 286 | 298
  Week 84 | 17.70 (6.779) | 17.27 (6.440)
  Week 96: number analyzed (Participants) | 259 | 268
  Week 96 | 17.24 (6.510) | 17.28 (6.480)
  Week 108: number analyzed (Participants) | 204 | 214
  Week 108 | 17.60 (6.580) | 17.07 (6.126)
  Week 120: number analyzed (Participants) | 148 | 158
  Week 120 | 18.18 (7.293) | 17.17 (6.416)
  Week 132: number analyzed (Participants) | 99 | 111
  Week 132 | 18.71 (7.926) | 16.52 (5.407)
  Week 144: number analyzed (Participants) | 65 | 74
  Week 144 | 18.02 (6.653) | 16.47 (6.805)
  Week 156: number analyzed (Participants) | 42 | 51
  Week 156 | 17.59 (5.937) | 17.21 (7.081)
  Week 168: number analyzed (Participants) | 21 | 28
  Week 168 | 16.60 (5.946) | 18.00 (8.052)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 15.52 (4.696) | 15.17 (7.808)
  Week 192: number analyzed (Participants) | 3 | 4
  Week 192 | 14.00 (3.568) | 16.45 (5.341)
  Early Term/Discontinuation: number analyzed (Participants) | 136 | 131
  Early Term/Discontinuation | 15.72 (5.512) | 15.58 (6.200)
  Final Visit: number analyzed (Participants) | 198 | 215
  Final Visit | 17.14 (7.356) | 16.03 (5.606)

8. Secondary Outcome: Vitamin K Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 441.826 Days), Final Visit (Mean: 946.463 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
ng/mL
  Baseline: number analyzed (Participants) | 443 | 429
  Baseline | 0.711 (0.6276) | 0.721 (0.6308)
  Week 12: number analyzed (Participants) | 410 | 393
  Week 12 | 0.752 (0.6601) | 0.769 (0.6887)
  Week 24: number analyzed (Participants) | 370 | 365
  Week 24 | 0.705 (0.6006) | 0.706 (0.6238)
  Week 36: number analyzed (Participants) | 337 | 350
  Week 36 | 0.739 (0.6726) | 0.748 (0.6630)
  Week 48: number analyzed (Participants) | 334 | 328
  Week 48 | 0.763 (0.6630) | 0.704 (0.6491)
  Week 60: number analyzed (Participants) | 322 | 330
  Week 60 | 0.761 (0.6868) | 0.778 (0.7247)
  Week 72: number analyzed (Participants) | 288 | 298
  Week 72 | 0.823 (0.7291) | 0.722 (0.6489)
  Week 84: number analyzed (Participants) | 273 | 283
  Week 84 | 0.780 (0.7174) | 0.725 (0.6869)
  Week 96: number analyzed (Participants) | 252 | 248
  Week 96 | 0.809 (0.7156) | 0.768 (0.6867)
  Week 108: number analyzed (Participants) | 191 | 201
  Week 108 | 0.802 (0.6797) | 0.768 (0.7119)
  Week 120: number analyzed (Participants) | 142 | 146
  Week 120 | 0.768 (0.6708) | 0.814 (0.7119)
  Week 132: number analyzed (Participants) | 93 | 104
  Week 132 | 0.824 (0.7655) | 0.760 (0.5740)
  Week 144: number analyzed (Participants) | 60 | 68
  Week 144 | 0.882 (0.7630) | 0.780 (0.6052)
  Week 156: number analyzed (Participants) | 40 | 50
  Week 156 | 0.754 (0.6129) | 0.816 (0.6822)
  Week 168: number analyzed (Participants) | 20 | 28
  Week 168 | 0.858 (0.6494) | 1.031 (0.8805)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 0.850 (0.7162) | 0.970 (0.9033)
  Early Term/Discontinuation: number analyzed (Participants) | 122 | 120
  Early Term/Discontinuation | 0.735 (0.7523) | 0.686 (0.5772)
  Final Visit: number analyzed (Participants) | 185 | 202
  Final Visit | 0.971 (0.7657) | 0.844 (0.6784)

9. Secondary Outcome: Serum Folate Levels
Time Frame: Baseline, Week 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 132, 144, 156, 168, 180, Early Term/Discontinuation (Mean: 423.024 Days), Final Visit (Mean: 946.074 Days)
Population: Safety population. This analysis was performed using the data only from patients who had the data at each visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AST-120 | Placebo
Number analyzed (Participants) | 507 | 509
ng/mL
  Baseline: number analyzed (Participants) | 489 | 487
  Baseline | 21.70 (44.420) | 21.78 (47.064)
  Week 12: number analyzed (Participants) | 452 | 450
  Week 12 | 21.47 (46.801) | 20.94 (45.093)
  Week 24: number analyzed (Participants) | 415 | 417
  Week 24 | 18.16 (34.095) | 19.46 (45.178)
  Week 36: number analyzed (Participants) | 382 | 383
  Week 36 | 20.95 (47.528) | 18.54 (41.653)
  Week 48: number analyzed (Participants) | 354 | 347
  Week 48 | 19.30 (44.798) | 21.50 (49.944)
  Week 60: number analyzed (Participants) | 322 | 333
  Week 60 | 19.06 (41.799) | 19.72 (45.119)
  Week 72: number analyzed (Participants) | 295 | 304
  Week 72 | 16.12 (32.761) | 19.96 (43.951)
  Week 84: number analyzed (Participants) | 271 | 288
  Week 84 | 17.00 (30.020) | 20.95 (46.184)
  Week 96: number analyzed (Participants) | 249 | 257
  Week 96 | 14.47 (25.918) | 18.17 (36.846)
  Week 108: number analyzed (Participants) | 192 | 199
  Week 108 | 13.50 (18.491) | 19.22 (39.625)
  Week 120: number analyzed (Participants) | 139 | 152
  Week 120 | 12.52 (16.033) | 17.01 (36.733)
  Week 132: number analyzed (Participants) | 94 | 105
  Week 132 | 17.09 (45.645) | 18.85 (44.240)
  Week 144: number analyzed (Participants) | 59 | 72
  Week 144 | 18.13 (41.386) | 18.09 (39.002)
  Week 156: number analyzed (Participants) | 40 | 49
  Week 156 | 13.08 (13.098) | 15.13 (20.162)
  Week 168: number analyzed (Participants) | 20 | 27
  Week 168 | 15.13 (12.776) | 16.26 (19.734)
  Week 180: number analyzed (Participants) | 6 | 12
  Week 180 | 33.10 (19.021) | 22.23 (25.137)
  Early Term/Discontinuation: number analyzed (Participants) | 129 | 121
  Early Term/Discontinuation | 24.43 (49.342) | 17.14 (24.122)
  Final Visit: number analyzed (Participants) | 192 | 214
  Final Visit | 15.52 (26.263) | 22.66 (50.498)

ADVERSE EVENTS:
Description: The AE analysis is based on the Safety Population. The Safety Population included all patients who were randomized and received at least 1 dose of study drug. The start number of Participant Flow included all patients who were randomized.
Arm/Group | AST-120 | Placebo
Serious Adverse Events (participants affected / at risk) | 195/507 | 184/509
Other Adverse Events (participants affected / at risk) | 376/507 | 382/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AST-120 (N=507) | Placebo (N=509)
Anaemia (Blood and lymphatic system disorders) | 8 | 7
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 5 | 3
Acute myocardial infarction (Cardiac disorders) | 7 | 5
Angina pectoris (Cardiac disorders) | 5 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 3 | 4
Cardiac failure acute (Cardiac disorders) | 1 | 3
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 11 | 9
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 3 | 5
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 5 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 2 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Open angle glaucoma (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 4
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Asthenia (General disorders) | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Catheter site related reaction (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 0 | 1
Lipogranuloma (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Appendicitis perforated (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Catheter site cellulitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 3
Cholecystitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 4
Gastroenteritis viral (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 2
Localised infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 2
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 13 | 13
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia herpes viral (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2
Pyelonephritis chronic (Infections and infestations) | 1 | 3
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 4
Urosepsis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 3 | 0
Blood glucose increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1
Diabetic foot (Metabolism and nutrition disorders) | 2 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 4
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Benign duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testicular seminoma (pure) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 3
Complex partial seizures (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 3
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Uraemic encephalopathy (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 4 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1
Glomerulonephritis acute (Renal and urinary disorders) | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 2
Renal failure acute (Renal and urinary disorders) | 9 | 22
Renal failure chronic (Renal and urinary disorders) | 48 | 45
Renal impairment (Renal and urinary disorders) | 3 | 3
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 2
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 16 | 8
Arteriovenous shunt operation (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Catheter placement (Surgical and medical procedures) | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 2 | 0
Dialysis device insertion (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Insertion of ambulatory peritoneal catheter (Surgical and medical procedures) | 2 | 6
Leg amputation (Surgical and medical procedures) | 0 | 1
Prosthesis implantation (Surgical and medical procedures) | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial stenosis (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypertensive crisis (Vascular disorders) | 5 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 3
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AST-120 (N=507) | Placebo (N=509)
Anaemia (Blood and lymphatic system disorders) | 58 | 81
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 | 5
Angina pectoris (Cardiac disorders) | 9 | 2
Bradycardia (Cardiac disorders) | 4 | 8
Hyperparathyroidism (Endocrine disorders) | 9 | 10
Hyperparathyroidism secondary (Endocrine disorders) | 11 | 17
Cataract (Eye disorders) | 14 | 9
Abdominal distension (Gastrointestinal disorders) | 13 | 10
Abdominal pain (Gastrointestinal disorders) | 11 | 15
Abdominal pain upper (Gastrointestinal disorders) | 13 | 6
Constipation (Gastrointestinal disorders) | 42 | 37
Diarrhoea (Gastrointestinal disorders) | 29 | 37
Dyspepsia (Gastrointestinal disorders) | 12 | 14
Faeces discoloured (Gastrointestinal disorders) | 1 | 6
Flatulence (Gastrointestinal disorders) | 7 | 12
Gastritis (Gastrointestinal disorders) | 6 | 14
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 8
Nausea (Gastrointestinal disorders) | 47 | 42
Vomiting (Gastrointestinal disorders) | 23 | 21
Asthenia (General disorders) | 17 | 11
Fatigue (General disorders) | 16 | 24
Oedema (General disorders) | 13 | 9
Oedema peripheral (General disorders) | 57 | 50
Pyrexia (General disorders) | 6 | 8
Seasonal allergy (Immune system disorders) | 2 | 6
Bronchitis (Infections and infestations) | 23 | 16
Cellulitis (Infections and infestations) | 7 | 2
Erysipelas (Infections and infestations) | 6 | 1
Gastroenteritis (Infections and infestations) | 13 | 9
Herpes zoster (Infections and infestations) | 3 | 6
Influenza (Infections and infestations) | 20 | 21
Nasopharyngitis (Infections and infestations) | 18 | 17
Pharyngitis (Infections and infestations) | 8 | 9
Pneumonia (Infections and infestations) | 4 | 9
Pyelonephritis chronic (Infections and infestations) | 3 | 8
Respiratory tract infection (Infections and infestations) | 16 | 12
Rhinitis (Infections and infestations) | 5 | 6
Sinusitis (Infections and infestations) | 7 | 12
Upper respiratory tract infection (Infections and infestations) | 24 | 31
Urinary tract infection (Infections and infestations) | 37 | 19
Ligament sprain (Injury, poisoning and procedural complications) | 6 | 1
Blood creatine phosphokinase increased (Investigations) | 10 | 8
Vitamin D decreased (Investigations) | 6 | 6
Acidosis (Metabolism and nutrition disorders) | 4 | 7
Decreased appetite (Metabolism and nutrition disorders) | 11 | 12
Dehydration (Metabolism and nutrition disorders) | 4 | 7
Dyslipidaemia (Metabolism and nutrition disorders) | 9 | 9
Fluid overload (Metabolism and nutrition disorders) | 7 | 1
Gout (Metabolism and nutrition disorders) | 24 | 21
Hypercalcaemia (Metabolism and nutrition disorders) | 8 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 35 | 36
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 21 | 26
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 14
Metabolic acidosis (Metabolism and nutrition disorders) | 18 | 27
Vitamin D deficiency (Metabolism and nutrition disorders) | 11 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 22
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 18
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 12
Dizziness (Nervous system disorders) | 8 | 11
Headache (Nervous system disorders) | 21 | 12
Depression (Psychiatric disorders) | 6 | 5
Insomnia (Psychiatric disorders) | 8 | 10
Renal failure acute (Renal and urinary disorders) | 5 | 8
Renal failure chronic (Renal and urinary disorders) | 42 | 55
Renal impairment (Renal and urinary disorders) | 10 | 6
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 21
Rash (Skin and subcutaneous tissue disorders) | 7 | 8
Arteriovenous fistula operation (Surgical and medical procedures) | 19 | 22
Hypertension (Vascular disorders) | 55 | 47
Hypotension (Vascular disorders) | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other